CLINICAL TRIAL: NCT06337500
Title: Validation of a Making Decision Hybrid (Ecologic and Virtual) Task
Acronym: LABLife
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023/764
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers; Behavior and Behavior Mechanisms
Keywords: decision-making; ecological task; brain activity
MeSH Terms: conditions — Behavior | interventions — Electroencephalography; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Iowa Gambling Task - ecologic (Experimental): The participant performs the card selection task in its ecological version (with real cards).
  Interventions: Other: Survey
- Iowa Gambling Task - virtual (Active Comparator): The participant performs the card selection task in its virtual version (computer task).
  Interventions: Device: Neurophysiological measure (EEG); Other: Survey
- Iowa Gambling Task - hybrid (Experimental): The participant performs the card selection task thanks to our homemade interface "LAB-Life".
  Interventions: Device: Neurophysiological measure (EEG); Other: Survey
- Game of Dice Task - ecologic (Experimental): The participant performs the dice-rolling task in its ecological version (with real dices).
  Interventions: Other: Survey
- Game of Dice Task - virtual (Active Comparator): The participant performs the dice-rolling task in its virtual version (computer task)
  Interventions: Device: Neurophysiological measure (EEG); Other: Survey
- Game of Dice Task - hybrid (Experimental): The participant performs the dice-rolling task thanks to our homemade interface "LAB-Life".
  Interventions: Device: Neurophysiological measure (EEG); Other: Survey

INTERVENTIONS:
Device: Neurophysiological measure (EEG) — Cerebral electric activity recorded with EEG
  Arms: Game of Dice Task - hybrid; Game of Dice Task - virtual; Iowa Gambling Task - hybrid; Iowa Gambling Task - virtual
Other: Survey — Participants complete a survey to evaluate their exposure to screens and their assessment of the laboratory task performed

SUMMARY:
The aim of this study is to validate a new hybrid (ecological + virtual) decision-making tool. The difference in behavior (risky choices) between the "hybrid" task and the "virtual" task will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 65 inclusive
* Subjects with no neurological or psychiatric disorders
* Subjects with no addictive disorder except tobacco
* Signed informed consent indicating that the subject has understood the purpose and procedures of the study and agrees to participate in the study and to abide by the requirements and restrictions inherent in the study
* Affiliation with a French social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Men and women under 18 or over 65 years of age
* Subjects suffering from a neurological or psychiatric disorder
* Subjects suffering from an addictive disorder, with the exception of tobacco
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator
* Subject without health insurance
* Pregnant
* Subject within the exclusion period of another study or on the "national volunteer list".

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Validation of the homemade "Lab-Life" interface as a tool for simulating an ecological task with sufficient fidelity, while meeting the conditions required for recording high-quality brain activity using an EEG-HR. | Day 1
  Behavioral score obtained after completion of the hybrid task (netscore obtained at the IGT). This score can be compared with the scores obtained after the ecological and virtual tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Julie GIUSTINIANI, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, Not in US/Canada, France

IPD SHARING:
Plan to Share IPD: No